CLINICAL TRIAL: NCT02870634
Title: A Phase 1 Single and Multiple Dose Escalation and Pharmacokinetic Study of Cu(II)ATSM Administered Orally to Patients With Amyotrophic Lateral Sclerosis/Motor Neuron Disease
Brief Title: Phase 1 Dose Escalation and PK Study of Cu(II)ATSM in ALS/MND
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Collaborative Medicinal Development Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMD-2016-001
Record Dates: First submitted 2016-08-10; First posted 2016-08-17 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Amyotrophic Lateral Sclerosis; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — copper (II) diacetyl-di(N(4)-methylthiosemicarbazone); Copper

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cu(II)ATSM (Experimental): Cu(II)ATSM capsules, administered orally once daily
  Interventions: Drug: Cu(II)ATSM

INTERVENTIONS:
Drug: Cu(II)ATSM — copper-containing synthetic small molecule
  Other Names: diacetylbis(N(4)-methylthiosemicarbazonato) copper(II)

SUMMARY:
Multicenter, open-label , single and multiple dose-escalation and pharmacokinetic study

DETAILED DESCRIPTION:
Multicenter, open-label, phase 1 study of Cu(II)ATSM administered orally to patients wit amyotrophic lateral sclerosis/motor neuron disease. The study will be conducted in three phases. In the first two phases, dose cohorts of six patients each will participate in a single dose pharmacokinetic study followed by a 28-day repeated daily dose study to establish the recommended phase 2 dose (RP2D). The first dose cohort will be treated at 3 mg/day; planned dose escalations are 6, 12, 24, and 48 mg/day, subject to observed safety assessments. In the third phase of the study, participants will be treated at the RP2D to confirm tolerability and assess preliminary evidence of efficacy.

In both the dose escalation and expansion cohorts, once the first 28 days of treatment and assessments are completed, at the discretion of the investigator a patient may continue to receive Cu(II)ATSM treatment for a maximum of six 28-day treatment cycles.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to initiation of any study-specific procedures;
* Familial or sporadic ALS/MND defined as clinically possible, probable, or definite by Awaji-shima Consensus Recommendations;
* First ALS/MND symptoms occurred no more than 2 years prior to screening visit;
* Seated FVC ≥ 70% and SNP ≥ 50% of predicted value;
* Not taking riluzole or on a stable dose of riluzole for at least 4 weeks prior to screening visit (participants are not allowed to start taking riluzole during the study);
* Age between 18 and 75 years at time of informed consent;
* Patient has a competent caregiver who can and will be responsible for administration of study drug;
* Adequate bone marrow reserve, renal and liver function:

  * absolute neutrophil count ≥ 1500/µL
  * lymphocyte count < 48%
  * platelet count ≥ 150,000/µL
  * hemoglobin ≥ 11 g/dL
  * creatinine clearance ≥ 60 mL/min (Cockroft & Gault formula)
  * ALT and/or AST ≤ 2 x ULN
  * total bilirubin ≤ 1.5 x ULN
  * serum albumin ≥ 2.8 g/dL
* Women and men with partners of childbearing potential must take effective contraception while on study and women of childbearing potential must have a negative pregnancy test and be non-lactating at screening

Exclusion Criteria:

* Inability to swallow oral medications or presence of GI disorder deemed to jeopardize intestinal absorption of Cu(II)ATSM
* Dependence of mechanical ventilation (non-invasive or invasive) for any part of day or night
* Exposure to any other investigational agent within 3 months or two investigational agents within 6 months prior to screening visit
* Active GI disease (except gastrointestingal reflux disease) within 30 days of screening visit
* Known immune compromising illness or treatment
* Presence of any of the following clinical conditions

  * drug abuse or alcoholism
  * unstable cardiac, pulmonary, renal, hepatic, endocrine or hematologic disorder
  * active infectious disease
  * AIDS or AIDS-related complex
  * current malignancy
  * unstable psychiatric illness, defined as psychosis or untreated major depression within 90 days of screening visit
  * neuromuscular disease other than ALS/MND
* Dementia that may affect either outcome measures or patient understanding and/or compliance with study requirements and procedures
* Use of anticoagulants at therapeutic doses within 7 days prior to screening visit
* Current use of strong inducers or inhibitors of CYPs 2C19 and 2D6

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-11-16 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
recommended phase 2 dose as determined by the number of participants at each dose level with dose limiting toxicities | 24 months

SECONDARY OUTCOMES:
Treatment-related change in disease severity by ALS Functional Rating Scale - Revised (ALSFRS-R) | 24 months
Treatment-related change in cognitive function by Edinburgh Cognitive and Behavioral Assessment (ECAS) score | 24 months
Treatment-related change in respiratory function by seated forced vital capacity (FCV) | 24 months
Treatment-related change in quality of life by ALSSQOL-R score | 24 months
Treatment-related change in disease severity by transcranial magnetic stimulation (TMS) response | 24 months
Peak Cu(II)ATSM plasma concentration following administration of a single dose based on blood draws taken at 1, 2, 4, 8 and 24 hours after dosing | 12 months
Area under the Cu(II)ATSM plasma concentration versus time curve (AUC) following administration of a single dose based on blood draws taken at 1, 2, 4, 8 and 24 hours after dosing | 12 months
Treatment-related change in respiratory function by sniff nasal pressure (SNP) test | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Rowe, MD, Principal Investigator — Macquarie University
Locations (2):
- Australia (2):
  - Macquarie University, Sydenham, New South Wales
  - Calvary Health Care Bethlehem, Caulfield, Victoria

IPD SHARING:
Plan to Share IPD: Undecided